CLINICAL TRIAL: NCT04637555
Title: A Multicenter Study to Evaluate the Long-term Safety and Tolerability of Open-label LCZ696 in Patients With Acute Myocardial Infarction Who Previously Participated in CLCZ696G2301 (PARADISE-MI)
Brief Title: Open-label Extension Study for CLCZ696G2301 (PARADISE-MI)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: CLCZ696G2301E1 extension study did not start as the core study (CLCZ696G2301) did not meet the primary endpoint.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696G2301E1; 2020-003906-29 (EudraCT Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Post Myocardial Infarction
Keywords: LCZ696; Open-Label Extension; PARADISE-MI; Post Myocardial Infarction; Post Heart Attack; CLCZ696G2301
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label extension study following-up to PARADISE-MI, which evaluated the efficacy and safety of LCZ696 compared to ramipril, in reducing the occurrence of CV death, heart failure (HF) hospitalization and outpatient HF (time-to-first event analysis) in post-acute myocardial infarction (AMI) patients with evidence of left ventricular (LV) systolic dysfunction and/or pulmonary congestion, without a known prior history of chronic HF. The study duration is up to approximately 24 months with visits at Days -14 to 1, 1, 15, 29 and Months 3, 6, 12, 18, and 24. Participants will receive LCZ696 at maximally tolerated doses with a target dose of 200 mg twice daily at all visits between day 1 and the last visit.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LCZ696 (sacubitril/valsartan) (Experimental): Following start of treatment, patients will receive LCZ696. Possible doses are level 1, 2, and 3 (50, 100 and 200 mg twice daily respectively)
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — LCZ696 (sacubitril/valsartan) tablet will be available in 24/26 mg, 49/51 mg and 97/103 mg, respectively
  Other Names: LCZ696

SUMMARY:
The purpose of this study is to collect long-term safety and tolerability data of LCZ696 and to provide open-label LCZ696 to eligible participants who completed CLCZ696G2301 study (PARADISE-MI) if LCZ696 is shown to have a positive benefit-risk profile in comparison to ramipril in reducing risk of cardiovascular (CV) mortality and development of heart failure in participants enrolled in the PARADISE-MI study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Participant received study treatment (either in LCZ696 or ramipril treatment arm) in PARADISE-MI.
3. Participant is safe to be enrolled in the extension study and may benefit from the treatment of LCZ696 per investigator's clinical judgement.

Exclusion Criteria:

1. Participant with a known history of angioedema
2. History of hypersensitivity to the study drug or drugs of similar chemical classes or known intolerance or contraindications to study drug or drugs of similar chemical classes including ACE inhibitors, ARB or NEP inhibitors
3. Symptomatic hypotension at screening
4. Serum potassium > 5.2 mmol /L (or equivalent plasma potassium value) at screening
5. Known hepatic impairment (as evidenced by total bilirubin > 3.0 mg/dL or increased ammonia levels, if performed), or history of cirrhosis with evidence of portal hypertension such as esophageal varices
6. Pregnant or nursing women or women of child-bearing potential unless they are using highly effective methods of contraception
7. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-26 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AE(s) leading to permanent study drug discontinuation, temporary study drug interruption, or study drug dose adjustment will be reported and summarized | Up to 24 months
  Adverse events (AEs) leading to treatment changes including treatment discontinuation, interruption, and dose adjustment
Number of participants with Serious Adverse Events (SAEs) | Up to 24 months
  SAE(s) will be reported, and the number of participants with SAE(s) will be summarized
Vital signs (Blood Pressure and pulse) | Baseline and up to 24 months
  BP and pulse will be measured at every visit. The test values of Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg) and heart rate (rate/minute) as well as change from the baseline will be summarized by parameter, using number of observations, mean, standard deviation, median, minimum, and maximum

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com